CLINICAL TRIAL: NCT05528809
Title: Quantification and Characterization of Circulating Epithelial and Endothelial Cells in Gougerot-Sjögren Syndrome, Compared to Systemic Sclerosis
Acronym: CIRCEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0043
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Primary Gougerot-Sjögren Syndrome; Systemic Sclerosis, Diffuse
Keywords: Sjögren's syndrome; systemic sclerosis; progenitor cells; circulating endothelial cells; circulating epithelial cells; endothelium; epithelium; autoimmune diseases; connective tissue disorders
MeSH Terms: conditions — Scleroderma, Diffuse; Sjogren's Syndrome; Scleroderma, Systemic; Autoimmune Diseases; Connective Tissue Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This a single-center prospective comparative non-randomized cohort pilot study, with 2 parallel groups (experimental group : patients with Gougerot-Sjögren's syndrome and positive control group : patients with diffuse systemic scleroderma).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Patients with Gougerot-Sjögren's syndrome meeting American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) disease definitions
  Interventions: Other: Blood sampling
- Positive control group (Active Comparator): Patients with diffuse systemic scleroderma meeting American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) disease definitions
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — A blood sampling will be performed during the inclusion visit (day 0).

SUMMARY:
Primary Gougerot-Sjögren's syndrome is a systemic autoimmune disease belonging to the group of connectivities, whose physiopathology remains largely unknown. Quantification and characterization of epithelial and endothelial circulants in Gougerot-Sjögren's syndrome could reflect the intensity of the epithelial aggression, and thus possibly constitute a biomarker.

DETAILED DESCRIPTION:
Primary Gougerot-Sjögren's syndrome is a systemic autoimmune disease belonging to the group of connectivities.

The criteria for classification of the disease include dry syndrome, positive salivary gland biopsy and detection of anti-Sjögren's-syndrome-related antigen A (anti-SSA) and anti-Sjögren's-syndrome-related antigen B (anti-SSB) antibodies. The presence of antibodies is thus important for the diagnosis but not essential, because in some patients the salivary gland biopsy is positive and the antibodies are absent. Therefore, the identification of new biomarkers could be very useful to confirm the diagnosis of primary Gougerot-Sjögren's syndrome and to identify subgroups of patients.

The pathophysiology of the disease remains largely unknown. Currently, primary Gougerot-Sjögren's syndrome is thought to originate from inflammation of the epithelial tissue of the salivary glands. However, it is currently unknown whether this autoimmune epithelitis is accompanied by a contingent of circulating epithelial cells, the characterization of which might be accessible by liquid biopsy.

So far, the circulating epithelial cells that have been identified have been identified in the context of cancer: in this case they are called circulating tumor cells. Their detection during primary Gougerot-Sjögren's syndrome could reflect the intensity of epithelial aggression, and thus possibly constitute a biomarker.

In other connectivities, data on circulating cells have already been published. In systemic scleroderma, another connectivitis affecting mainly middle-aged women, circulating progenitor cells have already been detected and are thought to have the capacity to differentiate into endothelial cells, thus playing a potentially important role in the pathophysiology of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over the age of 18
* Written and signed consent by the participant and the investigator
* Affiliated person or beneficiary of the social security system
* Test group: patients with Gougerot-Sjögren's syndrome connectivitis meeting the ACR/EULAR classification criteria
* Positive control group: patients with diffuse systemic scleroderma connectivitis meeting ACR/EULAR classification criteria

Exclusion Criteria:

* Association of the two diseases in the same patient
* Progressive cancer
* Subject protected by law, under guardianship or curatorship
* Inability to give free and informed consent to participate in the study
* Withdrawal of consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Circulating epithelial cell detection rate | day 0
  Rate of patients with at least 1 circulating epithelial cell in the peripheral blood

SECONDARY OUTCOMES:
Number of circulating epithelial cells | day 0
Number of circulating epithelial cells expressing human epidermal growth factor receptor 2 (HER2) | day 0
Number of circulating epithelial and endothelial cells | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GUILPAIN, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No